CLINICAL TRIAL: NCT06262711
Title: A Crossover Pilot Study on the Effects of Vitamin C Supplementation on Skeletal Muscle in Older Women (VICS)
Brief Title: Effects of Vitamin C on Skeletal Muscle
Acronym: VICS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of East Anglia (Other)
Collaborators: The Norfolk and Norwich University Hospitals NHS Foundation Trust (Unknown); The Quadram Institute Clinical Research Facility (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 321917
Record Dates: First submitted 2024-02-05; First posted 2024-02-16 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2024-01

CONDITIONS: Healthy
Keywords: skeletal muscle; mitochondrial function; muscle strength; physical function; vitamin C
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Crossover Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double blind masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C, then Placebo (Experimental): Participants will first consume one 500mg vitamin C capsule daily for 6 weeks. After a 4-week washout period, participants will crossover and consume one placebo capsule daily for 6 weeks.
  Interventions: Dietary Supplement: Vitamin C; Dietary Supplement: Placebo
- Placebo, then Vitamin C (Experimental): Participants will first consume one placebo capsule daily for 6 weeks. After a 4-week washout period, participants will crossover and consume one 500mg vitamin C capsule daily for 6 weeks.
  Interventions: Dietary Supplement: Vitamin C; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C — Vitamin C 500mg hydroxypropyl methylcellulose (HPMC) capsules (Solgar UK).
Dietary Supplement: Placebo — Vitamin C-matched placebo capsule. Placebo capsules manufactured using hydroxypropyl methylcellulose (HPMC) capsules and microcrystalline cellulose (MCC).

SUMMARY:
As part of the ageing process muscles become weaker. One of the reasons for this is that mitochondria, the 'engines' that provide energy to fuel muscles, age and work less efficiently. Mitochondria are found in almost all cells in the human body. Mitochondria take in nutrients that are provided from food and break these down to create energy-rich compounds to fuel many different processes in the body. Muscles are loaded with mitochondria because they require a lot of energy. Mitochondria naturally produce small compounds called oxidants that can damage muscle cells and can cause inflammation. The cells in the body have a natural defence system to protect against oxidants, but when mitochondria age and become less efficient, the amount of oxidants that they produce can increase. These oxidants can damage muscles and the mitochondria themselves. Antioxidants, such as vitamin C, may help protect muscles from the damage caused by oxidants, and may help mitochondria work more efficiently. In this study, the investigators will explore whether vitamin C can help mitochondria work more efficiently, which may improve muscle strength, and help older people to remain mobile and independent for longer.

DETAILED DESCRIPTION:
The VICS study is a 16-week randomised, double-blind, placebo-controlled two-arm crossover pilot study conducted between the Norfolk and Norwich University Hospital (NNUH) and the Quadram Institute Clinical Research Facility (QI CRF) in Norwich, UK. Investigators are seeking women over the age of 65 years with low habitual fruit and vegetable consumption to determine whether vitamin C supplementation affects mitochondrial function, compared to a matched placebo. Participants will attend 3 clinical visits where investigators will assess skeletal muscle mitochondrial function and membrane turnover using 31-phosphorous magnetic resonance spectroscopy (31P MRS). Investigators will assess muscle strength (hand grip strength and knee extension strength) measured using handheld dynamometers, and physical function measured using the short physical performance battery (SPPB). Investigators will monitor blood levels of vitamin C and inflammatory markers, specifically high-sensitivity C-reactive protein (hs-CRP), interleukin-6 (IL-6) and tumour necrosis factor-α (TNF-α), and the collagen markers procollagen type-1 N-terminal propeptide (P1NP) and collagen type-1 cross-linked C telopeptide (CTX). Participants will consume one oral capsule daily (containing either 500mg vitamin C or a matched placebo) for the first 6-week intervention period, then, after a 4-week washout phase, participants will crossover and consume the other capsule daily for the second 6-week intervention period. Participants will be asked to complete a food frequency (dietary) questionnaire and physical activity questionnaire at each visit to monitor their physical activity levels and fruit and vegetable consumption.

ELIGIBILITY:
Inclusion Criteria:

* Female, aged 65 years or over
* Non-smoker (or ex-smoker for at least 1 year).
* Engages in less than 20 minutes of structured physical activity per week, including cycling.
* Able to provide informed consent.
* Able to understand basic instructions in English.
* Willing to take daily vitamin C or placebo capsules.

Exclusion Criteria:

* Consumes more than 3 fruits and vegetables per day, including fruit and vegetable juices.
* Consumes vitamin C containing supplements, polyphenols, or other antioxidants (e.g. resveratrol or coenzyme q10).
* Regularly takes anti-inflammatory drugs.
* Alcohol intake >14 units/week.
* Chronic clinical diseases (e.g., coronary artery/peripheral artery/cerebrovascular diseases, diabetes, chronic kidney disease requiring dialysis, diagnosed low renal function, neurological disorders or diseases that may affect motor/cognitive functions), except hypertension and hyperlipidaemia.
* History of kidney stones within the preceding 12 months.
* Contraindications for undergoing the MRI and exercise study procedures (e.g. major surgery, bilateral hip or knee replacement, non-MRI-compatible pacemaker or metal implants).
* Parallel participation in another research project that involves an intervention.
* Relation to, or co-habitation with, a member of the study team.
* Those who are part of the line manager/supervisory structure of the Chief Investigator.

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — Biological Females
Enrollment: 16 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Difference in skeletal muscle mitochondrial function between vitamin C and placebo groups. | Week: 6 and 16
  Comparison of skeletal muscle mitochondrial oxidative capacity (estimated from 31P MRS measured phosphocreatine recovery half-time) following 6 weeks of vitamin C supplementation or 6 weeks of placebo.

SECONDARY OUTCOMES:
Difference in skeletal muscle phosphomonoester to phosphodiester ratio (PME/PDE) between vitamin C and placebo groups. | Week: 6 and 16.
  Skeletal muscle phosphomonoester (PME) and phosphodiester (PDE) concentrations can be measured using 31P MRS, and reflect cell membrane synthesis and breakdown respectively. The signal amplitudes (in arbitrary units) of these two species will be combined to report the (unitless) PME/PDE ratio, which reflects cell membrane turnover and may be related to oxidative stress. Comparison of PME/PDE ratio following 6 weeks of vitamin C or 6 weeks of placebo.
Difference in knee extension strength between vitamin C and placebo groups. | Week: 6 and 16.
  Comparison of knee extension strength following 6 weeks of vitamin C or 6 weeks of placebo.
Difference in hand grip strength between vitamin C and placebo groups. | Week: 6 and 16.
  Comparison of hand grip strength following 6 weeks of vitamin C or 6 weeks of placebo.
Difference in Short Physical Performance Battery (SPPB) score between vitamin C and placebo groups. | Week: 6 and 16.
  The Short Physical Performance Battery (SPPB) assesses three components of physical performance: standing balance, gait speed and chair stands. Each of the three components is scored from 0 (worst possible performance) to 4 (best possible performance). Scores from each of the three components are then summed to provide an overall SPPB score ranging from 0 (worst performance) to 12 (best performance). Comparison of SPPB score following 6 weeks of vitamin C or 6 weeks of placebo.
Difference in plasma vitamin C between vitamin C and placebo groups. | Week: 6 and 16.
  Comparison of plasma vitamin C following 6 weeks of vitamin C or 6 weeks of placebo.
Difference in serum hs-CRP between vitamin C and placebo groups. | Week: 6 and 16.
  Comparison of serum hs-CRP following 6 weeks of vitamin C or 6 weeks of placebo.
Difference in serum IL-6 between vitamin C and placebo groups. | Week: 6 and 16.
  Comparison of serum IL-6 following 6 weeks of vitamin C or 6 weeks of placebo.
Difference in serum TNF-α between vitamin C and placebo groups. | Week: 6 and 16.
  Comparison of serum TNF-α following 6 weeks of vitamin C or 6 weeks of placebo.
Difference in plasma P1NP between vitamin C and placebo groups. | Week: 6 and 16.
  Comparison of plasma P1NP following 6 weeks of vitamin C or 6 weeks of placebo.
Difference in plasma CTX between vitamin C and placebo groups. | Week: 6 and 16.
  Comparison of plasma CTX following 6 weeks of vitamin C or 6 weeks of placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Max Yates, Principal Investigator — Norfolk and Norwich University Hospitals NHS Foundation Trust
Locations (1):
- University of East Anglia, Norwich, Norfolk, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data supporting the findings of this study will be made available by the authors to any qualified researcher upon reasonable request.
Time Frame: Data will be made available upon publication of the study results, and will be available for 10 years from the study end date.
Access Criteria: Data request must be made by a qualified researcher.